CLINICAL TRIAL: NCT06913205
Title: Comparison of Regional Block Techniques Used for Postoperative Pain Management in Laparoscopic Appendectomy in Children
Brief Title: Rectus Sheath Block and Local Wound Infiltration in Pediatric Laparoscopic Appendectomies
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Hande Gurbuz, Assoc. Prof. MD. PhD, Bursa City Hospital
Other Study IDs: 2011-KAEK-25 2021/08-20
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Appendectomy, Laparoscopic; Pediatric Anesthesia; Nerve Block/Methods; Regional Anesthesia; Acute Pain, Postoperative
Keywords: laparoscopic appendectomy; pediatric anesthesia; nerve blocks; regional anesthesia; acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rectus Sheath Block: Children undergoing laparoscopic appendectomy with rectus sheath blocks
- Local infiltration: Children undergoing laparoscopic appendectomy with local infiltration

SUMMARY:
Laparoscopic appendectomy surgeries are among the most commonly performed procedures in childhood. However, they are associated with moderate to severe postoperative pain. Regional nerve block techniques are recommended for postoperative pain management. This research compared the two most frequently used methods: rectus sheath block and local wound infiltration.

DETAILED DESCRIPTION:
Acute appendectomy surgeries are one of the most frequently performed surgeries in childhood. Minimally invasive (laparoscopic) surgical methods are recommended, especially in abdominal surgeries, due to rapid wound healing, rapid recovery, less bleeding, and shorter hospital stays compared to open surgery. In addition to all these advantages of laparoscopic surgeries, postoperative somatic pain is expected to be less compared to open surgeries due to the small incisions in the abdominal wall. However, when the pain severity of children who underwent laparoscopic appendectomy was evaluated using the pain scoring scale, it was seen that the median pain scores were ≥7 in 5% of the children (severe pain) and ≥4 in 25% (moderate pain). Clinical practice guidelines also recommend the use of regional anesthesia and analgesia methods as part of multimodal analgesia in the prevention of intraoperative and postoperative pain. We also routinely use regional anesthesia and analgesia methods successfully and effectively in our daily practices in our clinic.

Rectus sheath blocks, which are known to be effective in midline incisions, and local anesthetic infiltrations of the wound site, which do not require special technical knowledge about regional anesthesia, are routinely applied in our clinic in every case. Although both methods provide clinical benefits, it is unknown which one is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* Older than 8 years
* Younger than 18 years
* Minimal invasive appendectomy (3 port)
* Consent to participate

Exclusion Criteria:

* Younger than 8 years
* Older than 18 years
* Convert to open abdominal surgery
* Do not consent to participate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing laparoscopic appendectomy surgery in Bursa Yuksek Ihtisas Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | Postoperative first 24 hours.
  Total acetaminophen use in the first 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative first 24 hours.
  Pain scores will be evaluated in the postoperative period using the Wong-Baker Faces Pain Rating Scale, where zero is equivalent to no pain, and 10 indicates the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data sets used in this research may be made available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Hamill JK, Liley A, Hill AG. Rectus sheath block for laparoscopic appendicectomy: a randomized clinical trial. ANZ J Surg. 2015 Dec;85(12):951-6. doi: 10.1111/ans.12950. Epub 2015 Jan 12. PMID 25581711
- [Background] Liu Y, Seipel C, Lopez ME, Nuchtern JG, Brandt ML, Fallon SC, Manyang PA, Tjia IM, Baijal RG, Watcha MF. A retrospective study of multimodal analgesic treatment after laparoscopic appendectomy in children. Paediatr Anaesth. 2013 Dec;23(12):1187-92. doi: 10.1111/pan.12271. Epub 2013 Sep 25. PMID 24112856
- [Background] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060
- [Derived] Gurbuz H, Karasu D, Dogan AK, Kilicarslan N. Rectus sheath blocks for pediatric laparoscopic appendicectomy. BMC Anesthesiol. 2025 Sep 29;25(1):462. doi: 10.1186/s12871-025-03364-9. PMID 41023777